CLINICAL TRIAL: NCT03976999
Title: Development of a Prospective and Monocentric Cinical and Biological Database in Epithelial Ovarian Cancer, Fallopian Tube Cancer and Primitive Peritoneal Cancer
Brief Title: Development of a Cinical and Biological Database in Ovarian, Fallopian Tube and Peritoneal Cancers
Acronym: BCBOvaire
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICM-BDD2016/04; 2016-A01041-50 (Registry Identifier: N° ID RCB)
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Peritoneal Neoplasms
Keywords: Biological Specimen Banks; Cancer; Gynecology
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological collection (Experimental): For all the patients include in the studie :
  * Blood samples collected at different times : Before treatment (T1) , after chemotherapy (T2), after interval surgery (T3) and after cancer reccurence (T4)
  * Tissue samples (tumor tissue and healthy tissue) collected during the surgery
  In parallel to this biological collection, standardized clinical data will be entered into a database
  Interventions: Other: Biological collection

INTERVENTIONS:
Other: Biological collection — * Blood samples collected at different times : Before treatment (T1) , after chemotherapy (T2), after interval surgery (T3) and after cancer reccurence (T4)
  * Tissue samples (tumor tissue and healthy tissue) collected during the surgery

SUMMARY:
A Clinical and Biological Database will provide to the scientific community a collection of blood and tissues with clinical datas to improve knowledge about cancer and help to develope new cancer treatments. This database is specific to epithetial ovarian cancer, Fallopian tube cancer and Primitive peritoneal cancer.

DETAILED DESCRIPTION:
A Clinical and Biological Database is a collection of reliable, prospective and representative datas.

This collection, provided to the scientific community, will help to develope research programs such as :

* Cinicals and biological predictive factors of treatments response
* Identification of biological tumoral markers associate with survival
* Identification of prognosic factors after recidivism
* Diagnostics tests optimisation and follow-up from blood samples ( Circulating Tumor Cells (CTC) )
* Developing strong preclinical models. Those models would be later used to test alternative treatments and would help to identify new biomarkers

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Patient at the diagnosis of an epithelial ovarian cancer, or a fallopian tube caner or a primitive peritoneal cancer
* Patient eligible for, at least, one surgery and a chemotherapy
* Patient having given his informed, written and express consent

Exclusion Criteria:

* Patient not affiliated to a social protection scheme
* Pregnant and / or nursing women
* Subject under tutelage, curatorship or safeguard of justice
* Patient whose regular follow-up is impossible for psychological, familial, social or geographical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-07-05 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who gave their consent to participate in the study | Until the study completion : 3 years
  The proportion of patients who consent to participate in the study among the screened patients

CONTACTS AND LOCATIONS:
Overall Officials: COLOMBO Pierre-Emmanuel, M.D, Principal Investigator — ICM - Institut régional du Cancer Montpellier
Locations (1):
- ICM - Institut régional du Cancer Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Result] Bolton KL, Chenevix-Trench G, Goh C, Sadetzki S, Ramus SJ, Karlan BY, Lambrechts D, Despierre E, Barrowdale D, McGuffog L, Healey S, Easton DF, Sinilnikova O, Benitez J, Garcia MJ, Neuhausen S, Gail MH, Hartge P, Peock S, Frost D, Evans DG, Eeles R, Godwin AK, Daly MB, Kwong A, Ma ES, Lazaro C, Blanco I, Montagna M, D'Andrea E, Nicoletto MO, Johnatty SE, Kjaer SK, Jensen A, Hogdall E, Goode EL, Fridley BL, Loud JT, Greene MH, Mai PL, Chetrit A, Lubin F, Hirsh-Yechezkel G, Glendon G, Andrulis IL, Toland AE, Senter L, Gore ME, Gourley C, Michie CO, Song H, Tyrer J, Whittemore AS, McGuire V, Sieh W, Kristoffersson U, Olsson H, Borg A, Levine DA, Steele L, Beattie MS, Chan S, Nussbaum RL, Moysich KB, Gross J, Cass I, Walsh C, Li AJ, Leuchter R, Gordon O, Garcia-Closas M, Gayther SA, Chanock SJ, Antoniou AC, Pharoah PD; EMBRACE; kConFab Investigators; Cancer Genome Atlas Research Network. Association between BRCA1 and BRCA2 mutations and survival in women with invasive epithelial ovarian cancer. JAMA. 2012 Jan 25;307(4):382-90. doi: 10.1001/jama.2012.20. PMID 22274685
- [Result] Colombo PE, Fabbro M, Theillet C, Bibeau F, Rouanet P, Ray-Coquard I. Sensitivity and resistance to treatment in the primary management of epithelial ovarian cancer. Crit Rev Oncol Hematol. 2014 Feb;89(2):207-16. doi: 10.1016/j.critrevonc.2013.08.017. Epub 2013 Sep 8. PMID 24071502
- [Result] Yang D, Khan S, Sun Y, Hess K, Shmulevich I, Sood AK, Zhang W. Association of BRCA1 and BRCA2 mutations with survival, chemotherapy sensitivity, and gene mutator phenotype in patients with ovarian cancer. JAMA. 2011 Oct 12;306(14):1557-65. doi: 10.1001/jama.2011.1456. PMID 21990299